CLINICAL TRIAL: NCT00820794
Title: A Phase 1, Open-Label, Randomized, Cross-Over Study To Estimate The Effects Of PD 0332334 On Lithium Pharmacokinetics In Healthy Subjects
Brief Title: A Phase 1 Study To Estimate The Effects Of PD 0332334 On Lithium Pharmacokinetics In Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A5361034
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Generalized Anxiety Disease
Keywords: Drug-drug interaction, lithium, PD 0332334, pharmacokinetics
MeSH Terms: interventions — Lithium; imagabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1a (Experimental): Subjects are treated with single dose lithium first. Then after at least 7 day washout, the subjects start PD 0332334 treatment from day 1 to day 9. At day 4 of PD 0332334 treatment, single dose lithium is given to subjects.
  Interventions: Drug: Lithium; Drug: PD 0332334
- Cohort 1b (Experimental): Subjects are treated with PD 0332334 from day 1 to 9 and a single dose of lithium is given at day 4. After at least 7 day washout, the subjects are treated with single dose of lithium.
  Interventions: Drug: Lithium; Drug: PD 0332334

INTERVENTIONS:
Drug: Lithium — 300 mg lithium, oral, once initially and then again at day 4 of PD 0332334 treatment
  Arms: Cohort 1a
Drug: PD 0332334 — 225 mg q12h PD 0332334, oral, 9 days treatment
  Other Names: imagabalin
  Arms: Cohort 1a
Drug: Lithium — 300 mg lithium, oral, at day 4 of PD 0332334 treatment and after 7 day washout
  Arms: Cohort 1b
Drug: PD 0332334 — 225 mg q12h PD 0332334, oral, 9 days treatment
  Arms: Cohort 1b

SUMMARY:
The purpose of this study is to investigate if PD 0332334 affects the pharmacokinetics of lithium by co-administering both drugs to healthy adults.

DETAILED DESCRIPTION:
Additional Study Purpose Details: To investigate potential drug-drug interaction between PD 0332334 and lithium

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and/or females
* Age from 21 to 55 (inclusive)
* BMI ranges from 18 to 30 kg/m2

Exclusion Criteria:

* Previous participation in a PD 332334 study
* Pregnant or nursing females
* Hypersensitivity (allergic) to lithium, Neurontin (gabapentin), or Lyrica (pregabalin)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Lithium pharmacokinetic endpoints: area under curve from 0 to infinity (AUCinf), area under curve from 0 to last quantifiable concentration (AUClast), half-life (T1/2), and maximum serum concentration (Cmax). | 10 days
The nature, incidence, duration, and severity of adverse events; discontinuation due to adverse events; clinical safety lab; 12-lead ECG; and vital signs will be monitored in this study. | 10 days

SECONDARY OUTCOMES:
No Secondary Outcomes | No Secondary Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361034&StudyName=A%20Phase%201%20Study%20To%20Estimate%20The%20Effects%20Of%20PD%200332334%20On%20Lithium%20Pharmacokinetics%20In%20Healthy%20Subjects